CLINICAL TRIAL: NCT04092881
Title: Efficacy of Short Pulsed 1064 nm Nd-YAG Laser Versus 10600 nm Fractional CO2 Laser in Treatment of Striae Alba: A Randomized Clinical Trial
Brief Title: Efficacy of Short Pulsed 1064 nm Nd-YAG Laser Versus 10600 nm Fractional CO2 Laser in Treatment of Striae Alba
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Manal Bosseila, Professor of dermatology - cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Short Nd-YAG vs Fr.CO2 for SA
Record Dates: First submitted 2019-08-03; First posted 2019-09-17 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Striae Distensae; Striae; Albicantes; Striae Alba; Nd-YAG Laser; Fractional CO2 Laser; High Frequency Skin Ultrasound; Short Pulsed Nd-YAG; Carbon Dioxide Laser; Neodymium-Doped Yttrium Aluminum Garnet Laser
Keywords: Striae Distensae; Striae; Albicantes; Striae Alba; Nd-YAG Laser; Fractional CO2 Laser; High Frequency Skin Ultrasound; Short Pulsed Nd-YAG; Carbon Dioxide Laser; Neodymium-Doped Yttrium Aluminum Garnet Laser
MeSH Terms: conditions — Striae Distensae | interventions — Lasers

STUDY DESIGN:
Intervention Model Description: * Written informed consent is to be obtained from each participant.
  * Detailed history taking including onset, course, duration of the disease and received medications.
  * Serial digital photography before and after each session and three months after sessions.
  * Clinical assessment to determine the severity of SD using modified Davey's visual score.
  * Comparable sides of striae are randomly allocated to one of the treatment modalities in a randomized table technique.
  * Application of four laser sessions one month apart using short pulsed mode of 1064 nm Nd-YAG laser (Fotona XP® Accelera mode) for one side and 10600 nm ablative fractional CO2 laser (Deka SmartXide DOT®) on the other. Sessions are separated by one month interval plus three months for clinical follow up.
  * Assessment using high frequency skin ultrasound before session, before 4th session and 3 months after last session.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Comparable sides of striae are randomly allocated to one of the treatment modalities in a randomized table technique.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Short pulsed Nd-YAG laser treatment side (Active Comparator): Neodymium-Doped Yttrium Aluminum Garnet (Nd-YAG) (Fotona XP®) laser is a successful therapeutic modality and is characterized by its safe profile compared to other lasers.
  Short pulsed Nd-YAG laser (Fotona XP® Accelera mode) results in a non-ablative dermal heating with intact overlying epidermis which has shown a potential for dermal collagen remodeling in histological sections.
  Interventions: Device: Laser
- Fractional ablative CO2 laser treatment side (Active Comparator): Carbon dioxide (CO2) (Deka SmartXide DOT®) laser is one of the well-tolerated therapeutic modalities used for treatment of different skin disorders including striae alba.
  CO2 laser targets mainly water content in both epidermis and dermis causing vaporization of target cells.
  Fractional ablative CO2 laser creates columns of focal dermo-epidermal tissue loss known as (microablative columns) with thermal damage, hemostatic effect and incomplete coagulation of tissues. This ablation of dermal tissues (including collagen and elastin) has the potential for stimulation of new tissue formation in striae distensae.
  Interventions: Device: Laser

INTERVENTIONS:
Device: Laser — Application of four laser sessions one month apart using short pulsed mode of 1064 nm Nd-YAG laser (Fotona XP® - Accelera mode) using parameters (fluence 20-40 J/Cm2, pulse duration= 0.25 ms and spot size 3-5 mm) for one side.
  Other Names: Short pulsed Nd-YAG laser (Fotona XP® device - Accelera mode)
  Arms: Short pulsed Nd-YAG laser treatment side
Device: Laser — Application of four laser sessions one month apart (in the same day after Nd-YAG session) using 10600 nm ablative fractional CO2 laser (Deka SmartXide DOT®) using -parameters (fluence 17-20 J/Cm2, pulse duration 700-1000 µs, spacing 600-700 µm and stacking 1-2) on the other. Sessions are separated by one month interval plus three months for clinical follow up.
  Other Names: Fractional ablative CO2 laser (Deka SmartXide DOT® device)
  Arms: Fractional ablative CO2 laser treatment side

SUMMARY:
Striae alba is a clinical variant of striae distensae characterized by focal dermal collagen loss and thinning of elastic fibers. Carbon dioxide (CO2) laser is an ablative laser modality that ablates defective collagen and stimulates new collagen formation. Neodymium-Doped Yttrium Aluminum Garnet (Nd-YAG) laser is a non ablative modality that results in stimulation of collagen formation through dermal heating. High frequency skin ultrasound is a rapid and non-invasive tool for measurement f skin thickness and can be used for this purpose.

DETAILED DESCRIPTION:
Striae distensae (SD) are skin disorders characterized by linear parallel edematous plaques that evolve into atrophic depressions in areas of dermal damage. They commonly develop on sites of skin stretching including thighs, arms and gluteal areas in males and additionally breasts in females, abdomen in case of pregnant females or intertreginous sites in case of glucocorticoids therapy and cushing disease.

All result in pathological changes comprising early dermal edema and perivascular lymphocytic infiltrate (manifest clinically as striae rubra) and end by epidermal thinning, flattening of dermal papillae, thinning of dermal collagen bundles and abundance of abnormally thinned and branched elastic fibers (manifest clinically as striae alba).

Various preventative and active treatment modalities for SD which were proven beneficial included: topical therapeutics like topical retinoids, energy based devices like fractional radiofrequency (FRF) and light therapy including both non-coherent light like intense pulsed light therapy and coherent laser devices like fractional ablative CO2 laser and non-ablative Nd-YAG laser. However obtaining a single effective treatment is still a challenge especially in absence of randomized control studies for some modalities and low level of evidence (LOE) for others.

Fractional ablative CO2 laser creates columns of focal dermo-epidermal tissue loss known as (microablative columns) with thermal damage, hemostatic effect and incomplete coagulation of tissues. This ablation of dermal tissues (including collagen and elastin) has the potential for stimulation of new tissue formation in SD. The efficacy of fractional CO2 laser in treatment of striae alba was discussed in various studies. In a LOE 4 retrospective study involved 27 patients each received one session of fractional ablative CO2 laser (at 10 mJ using ultrapulsed deep FX mode with spot diameter 1-10 mm) ; (7.4%) of patients have shown (>75 %) improvement, (51.9%) have shown (51 - 75%) improvement, (33.3%) have shown (26 - 50%) improvement and (7.4%) have shown (<25%) improvement. Another comparative study between both fractional ablative CO2 laser and non-ablative Erbium-glass laser with LOE=2 conducted on 22 patients using three sessions with four weeks interval. Fractional CO2 laser parameters were set to (fluence = 40-50 mJ, 75-100 spots/Cm2 spot density and spot size = 8x8 mm in a static mode). Results have shown marked clinical improvement in 90.9% of patients from both modalities with no statistically significant difference between both. A third comparative study (LOE=2) between fractional CO2 laser, FRF and combination between both included 30 patients using (fluence=700-1000 mJ and 0.7 mm spot density) for the fractional CO2 laser. Clinical improvement was noticed in all three groups with best results for the combination group. This result was supported by histopathological evidence in the form of increased epidermal and collagen thickness in analysis of biopsies retrieved from two patients. A Fourth comparative study (LOE=2) between combination of fractional ablative CO2 laser and microneedle FRF versus only microneedle FRF conducted on six patients using five sessions with four weeks interval. Fractional CO2 was conducted using (fluence = 14-18J/Cm2 and ablation depth = 400-600 micrometers in ultrapulsed mode using two passes). A statistically significant better result was noticed in the combination group with overall greater reduction in mean surface area of SD pointing to an additive positive role for fractional CO2 laser. A fifth comparative study between fractional CO2 laser versus combination of topical glycolic acid and tretinoin (LOE=2) conducted on six patients through five sessions with two to four weeks interval. Fractional CO2 was set to (fluence = 14-18 J/Cm2 in ultrapulsed mode). Statistically significant better results were noticed in fractional CO2 laser group with reduction in mean surface area of SD.

Neodymium-Doped Yttrium Aluminum Garnet (Nd-YAG) laser is another successful therapeutic modality and is characterized by its safe profile compared to other lasers. Long pulsed Nd-YAG laser results in a non-ablative dermal heating with intact overlying epidermis which has shown a potential for dermal collagen remodeling in histological sections (14). El Saie and his colleagues compared the efficacy of two fluences (75 J/Cm2 and 100 J/Cm2) of Nd-YAG using (spot size = 5 mm, pulse duration = 15 ms and frequency = 1 Hz) in the treatment of SD (both striae alba and rubra patients). Improvement was noticed in both types of striae. However, patients with striae alba showed better improvement in the higher fluence group. Increased dermal collagen and elastin were supported by histopathological evidences for biopsies retrieved from six patients. Nevertheless, other studies pointed to higher effectiveness in cases of striae rubra than striae alba which suggests an additional role for Nd-YAG laser in targeting dermal vascular changes in SD.

There were no previous attempts for comparing fractional ablative CO2 laser and long pulsed non-ablative Nd-YAG laser for treatment of striae alba patients. In a recent systematic review, a LOE=2 comparative study was conducted between 2940nm Erbium - Yettrium Aluminum Garnet (Er-YAG) ablative laser and non-ablative 1064nm Nd-YAG laser for treatment of patient with striae alba. Each group received three sessions with four weeks interval. Parameters were set to (power= 3.2 J and spot size= 7mm in a short pulsed mode) for Er-YAG laser and (fluence= 50 J/Cm2, spot size= 50 ms and pulse duration = 50ms) for Nd-YAG laser. Both groups have shown poor results. Overall conclusion from systematic review was that ablative lasers as an option for treatment of SD were less well-tolerated by patients and results were more variable among studies than non-ablative lasers.

Clinical evaluation of patients shall be determined by Davey's modified score for the number and severity of the striae in the affected area, both before and after treatment to determine the degree of improvement or worsening.

Objective evaluation of the efficacy of different therapeutic modalities is highly important to determine the optimal management. High frequency skin ultrasound (HFSU) is a rapid and non-invasive tool for measurement of skin thickness and can be used for this purpose, It is an ultrasound-based apparatus that emits ultrasound waves through a transducer in high frequencies that vary according to the designated visualized structure or tissue. In skin, 18 MHz devices are used primarily for dermal component imaging and 50-100 MHz devices for epidermal component imaging. Using bimodal devices is a more advanced option for visualization of ultrastructures of the dermis like collagen, elastic fibers and dermal ground substance.

Statistical analysis shall be done after study completion to determine the significance of the outcome parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients with striae alba.
* Ages between 14 years - 50 years.
* Both sexes.
* Skin types I-IV
* Bilateral striae.

Exclusion Criteria:

* Patients with striae rubra, striae nigra, striae caerulea or striae atrophicans.
* History of diseases associated with SD (cushing disease or Marfan syndrome).
* History of drugs associated with development of SD (topical or systemic glucocorticoids, Indinavir or protease inhibitors).
* History of conditions with abnormal dermal connective tissue structure (Ehler-Danlos syndrome, cutis laxa, pseudoxanthoma elasticum, elastolysis, elastomas, hyaline fibromatosis, keloidal tendencies, skin atrophy, poikiloderma or anetoderma).
* Current state of pregnancy in female patients.
* Relative contraindications to laser therapy (photosensitive dermatoses or burns).
* History of any therapeutic procedure for striae in the past 6 months before enrollment in the study.
* History of conditions associated with dermal edema or lymphedema.

Ages: 14 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of the efficacy and therapeutic superiority of both laser machines by measuring both clinical improvement using modified Davey's score and visually by measuring different skin thickness planes using high frequency skin ultrasound | 20 - 24 months
  Assessment of the efficacy and therapeutic superiority of either 1064 nm Nd-YAG laser or 10600 nm fractional CO2 laser as treatment modalities for patients with striae alba guided by investigated dermal changes obtained by high frequency skin ultrasound machine, namely: dermal thickness, sub epidermal low echogenicity band thickness and epidermal thickness, both before and after treatment with both laser machines. Statistical analysis of outcome data shall be carried out to determine significance of efficacy of one laser modality over the other.

SECONDARY OUTCOMES:
Treating and improving lesions of striae alba for 25 patients included in the sample size using both laser machines, one on each side in a rate of one session per month for four months duration | 20 - 24 months
  Treating and improving lesions of striae alba for all of the 25 patients included in the sample using short pulsed 1064 nm Nd-YAG laser and 10600 nm fractional CO2 laser each on one side of the area affected, for four successive sessions with one month interval. The degree of improvement shall be determined through comparing modified Davey's score both before and after treatment sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Heba Abd El-Kader, MD, Study Chair — Lecturer of Dermatology, Cairo University; Manal A. Bosseila, MD, Principal Investigator — Professor of Dermatology, Cairo University; Khaled El Kaffas, MD, Study Chair — Associate Professor of Investigative Radiology, Department of Radiology, Cairo University; Omar M. El-Ghanam, MSc, Study Director — Dermatology Specialist
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mikes BA, Oakley AM, Patel BC. Striae Distensae. 2025 May 19. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK436005/ PMID 28613776
- [Background] Ross NA, Ho D, Fisher J, Mamalis A, Heilman E, Saedi N, Jagdeo J. Striae Distensae: Preventative and Therapeutic Modalities to Improve Aesthetic Appearance. Dermatol Surg. 2017 May;43(5):635-648. doi: 10.1097/DSS.0000000000001079. PMID 28375972
- [Background] Omi T, Numano K. The Role of the CO2 Laser and Fractional CO2 Laser in Dermatology. Laser Ther. 2014 Mar 27;23(1):49-60. doi: 10.5978/islsm.14-RE-01. PMID 24771971
- [Background] Aldahan AS, Shah VV, Mlacker S, Samarkandy S, Alsaidan M, Nouri K. Laser and Light Treatments for Striae Distensae: A Comprehensive Review of the Literature. Am J Clin Dermatol. 2016 Jun;17(3):239-56. doi: 10.1007/s40257-016-0182-8. PMID 26923916
- [Background] Lee SE, Kim JH, Lee SJ, Lee JE, Kang JM, Kim YK, Bang D, Cho SB. Treatment of striae distensae using an ablative 10,600-nm carbon dioxide fractional laser: a retrospective review of 27 participants. Dermatol Surg. 2010 Nov;36(11):1683-90. doi: 10.1111/j.1524-4725.2010.01719.x. Epub 2010 Sep 14. PMID 20840494
- [Background] Yang YJ, Lee GY. Treatment of Striae Distensae with Nonablative Fractional Laser versus Ablative CO(2) Fractional Laser: A Randomized Controlled Trial. Ann Dermatol. 2011 Nov;23(4):481-9. doi: 10.5021/ad.2011.23.4.481. Epub 2011 Nov 3. PMID 22148016
- [Background] Ryu HW, Kim SA, Jung HR, Ryoo YW, Lee KS, Cho JW. Clinical improvement of striae distensae in Korean patients using a combination of fractionated microneedle radiofrequency and fractional carbon dioxide laser. Dermatol Surg. 2013 Oct;39(10):1452-8. doi: 10.1111/dsu.12268. Epub 2013 Jul 29. PMID 23895146
- [Background] Fatemi Naeini F, Behfar S, Abtahi-Naeini B, Keyvan S, Pourazizi M. Promising Option for Treatment of Striae Alba: Fractionated Microneedle Radiofrequency in Combination with Fractional Carbon Dioxide Laser. Dermatol Res Pract. 2016;2016:2896345. doi: 10.1155/2016/2896345. Epub 2016 Mar 16. PMID 27069471
- [Background] Naein FF, Soghrati M. Fractional CO2 laser as an effective modality in treatment of striae alba in skin types III and IV. J Res Med Sci. 2012 Oct;17(10):928-33. PMID 23825991
- [Background] Gianfaldoni S, Tchernev G, Wollina U, Fioranelli M, Roccia MG, Gianfaldoni R, Lotti T. An Overview of Laser in Dermatology: The Past, the Present and ... the Future (?). Open Access Maced J Med Sci. 2017 Jul 23;5(4):526-530. doi: 10.3889/oamjms.2017.130. eCollection 2017 Jul 25. PMID 28785350
- [Background] Gungor S, Sayilgan T, Gokdemir G, Ozcan D. Evaluation of an ablative and non-ablative laser procedure in the treatment of striae distensae. Indian J Dermatol Venereol Leprol. 2014 Sep-Oct;80(5):409-12. doi: 10.4103/0378-6323.140296. PMID 25201840
- [Background] Elsaie ML, Hussein MS, Tawfik AA, Emam HM, Badawi MA, Fawzy MM, Shokeir HA. Comparison of the effectiveness of two fluences using long-pulsed Nd:YAG laser in the treatment of striae distensae. Histological and morphometric evaluation. Lasers Med Sci. 2016 Dec;31(9):1845-1853. doi: 10.1007/s10103-016-2060-2. Epub 2016 Sep 5. PMID 27595152
- [Background] Hague A, Bayat A. Therapeutic targets in the management of striae distensae: A systematic review. J Am Acad Dermatol. 2017 Sep;77(3):559-568.e18. doi: 10.1016/j.jaad.2017.02.048. Epub 2017 May 24. PMID 28551068
- [Background] Bleve M, Capra P, Pavanetto F, Perugini P. Ultrasound and 3D Skin Imaging: Methods to Evaluate Efficacy of Striae Distensae Treatment. Dermatol Res Pract. 2012;2012:673706. doi: 10.1155/2012/673706. Epub 2011 Nov 22. PMID 22203840
- [Background] Davey CM. Factors associated with the occurrence of striae gravidarum. J Obstet Gynaecol Br Commonw. 1972 Dec;79(12):1113-4. doi: 10.1111/j.1471-0528.1972.tb11896.x. No abstract available. PMID 4646568
- [Background] Al-Himdani S, Ud-Din S, Gilmore S, Bayat A. Striae distensae: a comprehensive review and evidence-based evaluation of prophylaxis and treatment. Br J Dermatol. 2014 Mar;170(3):527-47. doi: 10.1111/bjd.12681. PMID 24125059